CLINICAL TRIAL: NCT06009692
Title: Effects of Neuro-dynamic Mobilization Techniques on Upper Limb Functions in Pronator Teres Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Umaira Sattar
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pronator Teres Syndrome
Keywords: Upper limb functions; Neurodynamics; Pronator Teres Syndrome; Task Oriented training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Limb Neurodynamics Group (Experimental): Upper limb Neuro-dynamics (Slider/Tensioner Technique) along with Task Oriented Training
  Interventions: Other: Upper limb Neuro-dynamics (Slider/ Tensioner Technique)
- Upper Limb Conventional Therapy (Active Comparator): Stretching, Strengthening exercises along with Task Oriented Training
  Interventions: Other: Conventional Therapy for Upper limb

INTERVENTIONS:
Other: Upper limb Neuro-dynamics (Slider/ Tensioner Technique) — The experimental group will receive neuro-dynamic mobilization techniques along with task oriented training. Slider versus tensioner technique will be applied according to each patient's need. Session time will be 25-30 minutes. Four series of 10 tensioning movements at a rhythm of ∼6s per cycle and 1 min rest between each series will be performed. After each cycle of 10 repetitions, the position will hold for 10s.
  Arms: Upper Limb Neurodynamics Group
Other: Conventional Therapy for Upper limb — Conventional treatment will include therapeutic ultrasound for 4 min, TENS for 10 min. Task oriented training will be designed according to patient's functional outcomes. Sessions will be given for 6 days a week, 25-30 minutes per day.
  Arms: Upper Limb Conventional Therapy

SUMMARY:
The study aimed to determine the effects of neuro-dynamic techniques on upper limb motor and sensory functions and to compare the effects of slider versus tensioner neuro-dynamic techniques on upper limb motor and sensory functions in pronator teres syndrome.

DETAILED DESCRIPTION:
The study aimed to determine the effects of neuro-dynamic techniques on upper limb motor and sensory functions and to compare the effects of slider versus tensioner neuro-dynamic techniques on upper limb motor and sensory functions in pronator teres syndrome.

Pronator teres syndrome is a rare condition and easily overlooked and mistaken for the more prevalent carpal tunnel syndrome. The median nerve may also be squeezed between the heads of the pronator teres muscle in addition to the carpal tunnel. Patients report pain, numbness, or paresthesia over the lateral 3.5-digit area and anterior forearm, which worsens with forced pronation. This condition is most common in the dominant hand or sometimes can be associated with advanced forearm muscle.in our routine clinical practice, The neuro-dynamic techniques is not that common in neurological physical therapy practice so the effects of neuro -dynamics with conventional therapy needs to be evaluated for better outcomes in upper limb functions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pronator teres syndrome
* At least 6 working hours/ day
* Positive Tinel's sign at pronator area (Hoffman's sign)
* Positive Pronator teres syndrome test

Exclusion Criteria:

* Any previous history of metabolic disease, liver disease/ diabetes
* History of previous injuries to the cervical spine including radiculopathies and myelopathies as well as spinal stenosis and/or spinal disc herniation

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Numeric visual analogue scale (VAS) | 2 weeks
  Numeric visual analogue scale (VAS) is a self-reported assessment that consists of a line with severe anchors ranging from "no pain" to "intense pain", which can be vertical or horizontal. Most frequently 10 cm long, this line serves as a continuum of pain severity. High test-retest reliability for the VAS has been recorded (ICC = 0.71-0.99). VAS is regarded as a powerful, therapeutically practical, accurate, and true measure of pain severity.
Upper Extremity Functional Scale (UEFS) | 2 weeks
  Upper Extremity Functional Scale (UEFS) is an 8-item, region-specific questionnaire designed to evaluate diseases of the upper extremities caused by work. The UEFS is a valid, reliable, and responsive tool created to assess how patients with a range of diseases are affected by upper extremity disorders in terms of function. UEFS demonstrate good internal consistency (Cronbach alpha > 0.83).
Jamar hand held dynamometer | 2 weeks
  Jamar hand held dynamometer is widely used in clinical practice and research as a result of the American Society of Hand Therapists (ASHT) recommendation of it as the gold standard. The ICC for the Jamar dynamometer ranged from .996 to .998 (p< 0.05).
Range of Motion | 2 weeks
  Goniometer is a method for measuring joint range of motion (ROM) that is widely accepted. It uses accurate and reliable measurement tools, especially the universal goniometer. For goniometry, Intraclass Correlation Coefficients (ICC- 3, k) of 0.94 showed excellent intra-ratter reliability.
Nottingham sensory assessment Scale | 2 weeks
  The Nottingham sensory assessment is a standardized scale for assessing sensory assessment in stroke patients. The NSA consists of 20 items and four subscales. The subscales included proprioception, stereognosis, two-point discrimination and tactile feeling. Each subscales item on tactile location on both sides of the body and bilateral simultaneous contact can be graded on the scale of 0-2. The Cronbach's alpha was used to evaluate internal consistency, values over 0.70 indicate Strong internal consistency.
Wolf Motor Function Test | 2 weeks
  Wolf Motor Function Test (WMFT) quantifies upper extremity movement ability through timed single- or multiple-joint motions and functional tasks. The original version consisted of 21 item; the widely used version of the WMFT consists of 17 items Composed of 3 parts: Time, Functional ability &Strength. It Includes 15 function-based tasks and 2 strength based tasks Performance time is referred to as WMFT-TIME. Functional ability is referred to as WMFT-FAS. Items 1-6 involve timed functional tasks, items 7-14 are measures of strength, and the remaining 9 items consist of analyzing movement quality when completing various tasks. The WMFT is an instrument with high inter rater reliability, internal consistency, test-retest reliability, and adequate stability.

CONTACTS AND LOCATIONS:
Overall Officials: Abrish Habib Abbasi, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Al-Nafees hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No